CLINICAL TRIAL: NCT03225391
Title: Effect of Programmed Naps on Decision Making of Residents During Working Hours.
Brief Title: Effect of Naps on Decision Making of Residents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Armando Castorena-Maldonado, Head of Otolaryngology Department, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: C05-11
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Internship and Residency; Sleep; Decision Making
Keywords: Residents; Naps; decision making

STUDY DESIGN:
Who Masked: Investigator
Masking Description: At the moment of running the Iowa Gambling Task and the Psychomotor Visual Test the investigator does not know the schedule of the nap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nap 1 (Experimental): Subjects who take, during a night shift, first a nap from 0:00 to 3:00 hours and, after 6 weeks of lavage, another nap from 3:00 to 6:00 hours.
  Interventions: Behavioral: nap from 0:00 to 3:00 hours; Behavioral: nap from 3:00 to 6:00 hours
- Nap 2 (Experimental): Subjects who take, during a night shift, first a nap from 3:00 to 6:00 hours and, after 6 weeks of lavage, another nap from 0:00 to 3:00 hours.
  Interventions: Behavioral: nap from 0:00 to 3:00 hours; Behavioral: nap from 3:00 to 6:00 hours

INTERVENTIONS:
Behavioral: nap from 0:00 to 3:00 hours — A nap from 0:00 to 3:00 hours during a night shift.
Behavioral: nap from 3:00 to 6:00 hours — A nap from 3:00 to 6:00 hours during a night shift.

SUMMARY:
Sleep deprivation produces changes including alteration of mood, irritability, fatigue, less focus and disorientation, also perceptive distortions, visual hallucinations and considering tasks harder and less pleasant. In resident physicians, these alterations have been shown to affect their work performance. Naps have proved to improve arousal and attention, alertness and performance. Those longer than 90 minutes promote a learning process similar to that occurring in REM sleep. Therefore a nap schedule could improve the decision making of residents during their working hours.

DETAILED DESCRIPTION:
Sleep deprivation produces changes including alteration of mood, irritability, fatigue, less focus and disorientation, also perceptive distortions, visual hallucinations and considering tasks harder and less pleasant. Extenuating working hours provoke sleep deprivation, which deteriorates work performance, produces mood disorders and increase chances of error.

In a survey performed to 3600 resident physicians in the USA it was observed that working more than 24 continuous hours was related with a higher risk of traffic accidents, as well as a higher tendency towards medical mistakes due to overstress, the most common being a diminished capability of performing a previously known procedure; also there were difficulties to solve problems generated by coworkers or relatives. Other study determinated that after a night shift the levels of daytime sleepiness were similar or higher than those of patients with narcolepsy or sleep apnea. The lack of sleep affects the performance of tasks, producing alterations similar to those in alcoholic intoxication, with a decline in visual attention, reaction speed, visual memory and creative thinking. Even though the effects of sleep deprivation in resident have been difficult to quantify due to confounders, there are indicators as decline in performance, which seems higher in less experienced physicians, with a higher alteration in reasoning and reaction time. It has been found in physicians in training (anesthesiology residents) that mistakes in administration of epidural anesthesia are more frequent after sleep deprivation; and a resident performing monitoring tasks after a night shift was more liable to mistakes that after a resting night, being also less likely to recognize arrhythmias in an electrocardiogram. Sleep deprivation affects coordination and skill, as observed in laparoscopist surgeons who took more time to complete a procedure after sleep deprivation than those who had rested. This results made the ACGME to establish a limitation in working hours during the residence.

Naps from 30 minutes to 4 hours improve alertness and performance. Studies comparing naps and caffeine have shown that naps not only improve arousal and attention but also helps to consolidate memory in those longer than 90 minutes. Furthermore, naps with slow wave and REM sleep are partially equivalent to a night's sleep, restoring the damage from baseline. It has been proven that naps promote a learning process similar to that occurring in a complete night sleep, which correlates with phase 2 of REM sleep. Therefore a nap schedule could improve the decision making of residents during their working hours.

ELIGIBILITY:
Inclusion Criteria:

* Resident physician cursing the first to third year in the pulmonology or pediatric pulmonology residency of the INER.
* Accepts to participate in the study signing the informed consent.

Exclusion Criteria:

* Chronic-degenerative or psychiatric disease.
* Sleep disorders diagnosed before recruiting.

Elimination Criteria:

* Not performing all psychometric tests.
* Lack of data in questionnaire.

Ages: 23 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Decision making | At 12:00 on the day of the nap.
  Net total and demographically corrected percentile in the Iowa Gambling Task.

SECONDARY OUTCOMES:
Alertness | At 12:00 hours on the day of the nap.
  Mean reaction time in the psychomotor vigilance test.
Sleep quality | 3 hours.
  Sleep efficiency as assessed by actigraphy
Vigilance | At 12:00 hours on the day of the nap.
  Slope of the reaction time in the psychomotor vigilance test.
Energy Expenditure | 22 hours around the nap.
  Total activity kcal as calculated via algorithm by actigraphy.
Activity | 22 hours around the nap.
  Percentages of sedentary, light, vigorous and very vigorous activity as calculated via algorithm by actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Armando R Castorena-Maldonado, MD, Principal Investigator — Insituto Nacional de Enfermedades Respiratorias
Locations (1):
- Insituto Nacional de Enfermedades Respiratorias, Mexico City, Delegacion Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Halbach MM, Spann CO, Egan G. Effect of sleep deprivation on medical resident and student cognitive function: A prospective study. Am J Obstet Gynecol. 2003 May;188(5):1198-201. doi: 10.1067/mob.2003.306. PMID 12748477
- [Background] Rollinson DC, Rathlev NK, Moss M, Killiany R, Sassower KC, Auerbach S, Fish SS. The effects of consecutive night shifts on neuropsychological performance of interns in the emergency department: a pilot study. Ann Emerg Med. 2003 Mar;41(3):400-6. doi: 10.1067/mem.2003.77. PMID 12605209
- [Background] Schweitzer PK, Randazzo AC, Stone K, Erman M, Walsh JK. Laboratory and field studies of naps and caffeine as practical countermeasures for sleep-wake problems associated with night work. Sleep. 2006 Jan;29(1):39-50. doi: 10.1093/sleep/29.1.39. PMID 16453980
- [Background] Killgore WD, Balkin TJ, Wesensten NJ. Impaired decision making following 49 h of sleep deprivation. J Sleep Res. 2006 Mar;15(1):7-13. doi: 10.1111/j.1365-2869.2006.00487.x. PMID 16489997
- [Background] Mednick SC, Nakayama K, Cantero JL, Atienza M, Levin AA, Pathak N, Stickgold R. The restorative effect of naps on perceptual deterioration. Nat Neurosci. 2002 Jul;5(7):677-81. doi: 10.1038/nn864. PMID 12032542